CLINICAL TRIAL: NCT06951451
Title: Effect of Smartphone Application (MED-AD) on Medication Adherence Among Patients With Cardiovascular Disease in Oman: A Multicenter Randomized Clinical Trial
Brief Title: Effect of Smartphone Application (MED-AD) on Medication Adherence Among Patients With Cardiovascular Disease in Oman
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sultan Qaboos University (Other)
Responsible Party: Principal Investigator, Dr. Huda Al Noumani, Associate Professor, Department of Adult Health and Critical Care, Sultan Qaboos University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MoH/CSR/22/26909
Record Dates: First submitted 2025-04-20; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Ischemic Cardiovascular Disease; Hypertension; Hyperlipidemia
MeSH Terms: conditions — Hypertension; Hyperlipidemias

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MED-AD application (Experimental): MED-AD is a smartphone application that will use two strategies (pill reminders and educational notifications) to enhance medication adherence. Both methods have shown their effectiveness in independently improving medication adherence; however, combining two or more strategies maximizes the efficacy of improving adherence. In addition, this application will be unique as it allows the patient to engage with their self-management behaviors and get feedback about their performance. The research team will develop the smartphone application with an expert in the application development field. In addition, the research team will pilot the MED-AD application on the same population and modify it before implementation of the study. The application will be hosted on SQU's in-house data, which is hosted and managed by the Center for Information Systems.
  Interventions: Behavioral: smartphone application (MED-AD)
- Short Text-message Reminders (Active Comparator): Participants will receive short text messages (SMS) to remind them to take medications as prescribed once daily. However, unlike the application reminders, the SMS will be general and not specify taking particular medicines. An example of the SMS message will be, "Remember to take your medicines for the day?" The research team will pilot the MED-AD application on the same population and modify it before implementing the study.
  Interventions: Behavioral: Short Text-message Reminders
- Routine care (No Intervention): Participants will receive routine care that does not include text messages or reminders and education through an application. In primary health care centers, the current routine care for people with chronic disease consists of the physical attendance of patients to their pre-scheduled medical appointment. The medical appointment will be every three months for most regular and controlled cases. The health care provider will usually evaluate the patient's condition, including the disease progression and medication adherence, and compare that with clinical parameters and laboratory investigations. Medications will be prescribed for the next three months, but the dispensing will be monthly. Patients will come every month directly to the pharmacy for a medication refill. The pharmacist will check the time window for medication refills and dispense the prescribed medications for one month.

INTERVENTIONS:
Behavioral: smartphone application (MED-AD) — 1. Medication Reminders: The oral medication list of the patient (names, doses, times, and frequency of administration) will be entered manually in the application by the RA in agreement with the patient during the medication prescription refill. This application will then send reminders, as notifications and voice notes, to take medications. An example of the reminder is "take lisinopril, one tablet, 10 mg at 9:00 am." The reminders will be categorized as normal, urgent & critical. Normal is a reminder sent on the normal medication timing. An urgent reminder is when the patient misses confirming a reminder more than once, which will be set as an alert on the phone. Critical reminder is when the patient misses confirming a reminder multiple times, which will be as an alert or an alarm on the phone. In addition, the application will notify a family member in case of urgent and critical reminders.
  2. Medication Adherence Report: The application will generate a weekly report on medication
  Arms: MED-AD application
Behavioral: Short Text-message Reminders — Participants will receive short text message (SMS) reminders to remind them to take medications as prescribed ONCE daily. However, the SMS will be general and not specify taking particular medicine compared to the application reminders. An example of the SMS message will be "Remember to take your medicines of the day?" The research team will pilot the MED-AD application on the same population and modify it before the implementation of the study.
  Arms: Short Text-message Reminders

SUMMARY:
This study aims to:

1. Investigate the impact of MED-AD intervention on medication adherence among CVD patients, compared to patients receiving text message reminders or routine care alone at baseline, 6 months, and 12 months later.
2. Evaluate the effectiveness of MED-AD intervention on clinical outcomes among patients with CVD, compared to the outcomes of patients receiving text or routine care alone at baseline, 6 months, and 12 months later.

This study is a prospective randomized controlled clinical trial (RCT) with three arms:

1. MED-AD intervention: MED-AD is a smartphone application that will use the following strategies (pill reminders, Medication Adherence Report, medication intake confirmation, Medical Appointment Reminder, and educational notifications) to enhance medication adherence
2. Text message reminders: Participants will receive short text message (SMS) reminders to remind them to take medications as prescribed once daily
3. Routine care only: Participants will receive routine care that does not include text messages or reminders and education through an application.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosed with at least one CVD (i.e., HTN, IHD, hyperlipidemia),
2. prescribed at least one medication for at least one year,
3. Omanis aged 18 years or older,
4. registered in the selected healthcare center, and 5) agreed to participate in the study

Exclusion Criteria:

1. have a severe cognitive impairment,
2. are unable to provide informed consent,
3. cannot read, and 4) do not have a smartphone with a compatible operating system (ios or Android).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Adherence to Refills and Medications Scale | BASELINE, AT 6 MONTHS, AT 12 MONTHS
  This instrument includes 12 items divided into two subscales: 8 items on the medication-taking subscale and four items on the refill subscale. The items are scored on a 4-point Likert scale with ranges of 1 = ''none of the time'' to 4 = ''all of the time.'' The total score is the sum of all items, ranging from 12 to 48, with lower scores representing better medication adherence.
The Proportion of Days Covered | BASELINE, AT 6 MONTHS, AT 12 MONTHS
  This measure is one of the objective, indirect instruments used to measure adherence. It calculates the number of days "covered" over the total number of days in the same period.
  Proportion of days covered = Days Supply of medication dispensed to the patient/ Total number of days X 100%
  The scoring is always positive and ranges from 0 to 100%. Zero means no adherence, while a PDC of 100% indicates perfect adherence. The threshold is the level that provides a reasonable likelihood of achieving the clinical benefits of therapy. For patients with cardiovascular diseases (CVD), clinical evidence supports using 80% as a standard PDC threshold.

SECONDARY OUTCOMES:
Clinical outcomes | BASELINE, AT 6 MONTHS, AT 12 MONTHS
  laboratory findings (i.e., Blood pressure, Cholesterol level, triglyceride levels, LDL, HDL, Ejection fraction, GFR), and cardiovascular complications in the previous three months (i.e., heart failure, dysrhythmias, strokes, heart attacks, Catheterization, ED visits, hospitalization, LOS if hospitalized, cardiac enzymes[troponin I])

CONTACTS AND LOCATIONS:
Locations (1):
- Ministry of Health, Muscat, Oman

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: The study protocol will be made available upon reasonable request beginning 3 months after the primary results are published. Requests must include a methodologically sound proposal and will be subject to review.
Access Criteria: Qualified researchers affiliated with academic, healthcare, or research institutions can access the study protocol only; no individual participant data (IPD) will be shared. The protocol includes detailed information about the study design, objectives, and methodology. It will be made available upon reasonable request starting three months after publication of the primary study results. Access will be granted following a brief review process to ensure appropriate use, and the document will be shared through secure institutional email or document-sharing platforms.
URL: https://www.icmje.org/recommendations/browse/publishing-and-editorial-issues/clinical-trial-registration.html